CLINICAL TRIAL: NCT04296578
Title: A Phase 1 Study Evaluating the Efficacy and Safety of Sodium Selenite in Combination With Abiraterone in Patients With Castrate Resistant Prostate Cancer Progressing on Abiraterone
Brief Title: Study Evaluating Sodium Selenite in Combination With Abiraterone in Castrate Resistant Prostate Cancer Progressing on Abiraterone
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study did not start
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-52111; PROS0097 (Other: OnCore)
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer; Castrate Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Sodium Selenite; Prednisone

STUDY DESIGN:
Intervention Model Description: Dose-finding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: 5.5 mg selenite (Experimental): Given orally, 5.5 mg selenite with food (within 30 mins of eating), for 5 weeks and monthly there after
  Interventions: Drug: Abiraterone Acetate; Drug: Sodium Selenite; Drug: Prednisone
- Cohort 2: 11 mg selenite (Experimental): Given orally, 11 mg selenite with food (within 30 mins of eating) for 5 weeks and monthly there after
  Interventions: Drug: Abiraterone Acetate; Drug: Sodium Selenite; Drug: Prednisone
- Cohort 3: 16.5 mg selenite (Experimental): Given orally, 16.5 mg selenite with food (within 30 mins of eating) for 5 weeks and monthly there after
  Interventions: Drug: Abiraterone Acetate; Drug: Sodium Selenite; Drug: Prednisone
- Cohort 4: 22 mg selenite (Experimental): Given orally, 22 mg selenite with food (within 30 mins of eating) for 5 weeks and monthly there after
  Interventions: Drug: Abiraterone Acetate; Drug: Sodium Selenite; Drug: Prednisone
- Cohort 5: 27.5 mg selenite (Experimental): Given orally, 27.5 mg selenite with food (within 30 mins of eating) for 5 weeks and monthly there after
  Interventions: Drug: Abiraterone Acetate; Drug: Sodium Selenite; Drug: Prednisone
- Cohort 6: 33 mg selenite (Experimental): Given orally, 33 mg selenite with food (within 30 mins of eating) for 5 weeks and monthly there after
  Interventions: Drug: Abiraterone Acetate; Drug: Sodium Selenite; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Standard of Care (SOC) abiraterone (Zytiga) as per package insert. The recommended dose of ZYTIGA is 1,000 mg (four 250 mg tablets) administered orally once daily in combination with prednisone 5 mg administered orally twice daily.
  Other Names: Zytiga; Yonsa; CB7630
Drug: Sodium Selenite — 11 mg tablets
  Other Names: Sodium selenite pentahydrate
Drug: Prednisone — SOC prednisone 5 mg PO twice daily
  Other Names: 1, 2-dehydrocortisone; Prednisonum; deltacortisone; deltadehydrocortisone

SUMMARY:
The purpose of this study is to access the safety of combining sodium selenite with abiraterone and to see what doses of sodium selenite can be safely combined with abiraterone in treating castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE(S):

· To determine the maximum tolerated dose (MTD) of sodium selenite when given in combination with abiraterone.

SECONDARY OBJECTIVE(S):

* To assess the safety and tolerability of the combination of sodium selenite and abiraterone in subjects with castration resistant prostate cancer (CRPC)
* To assess the pharmacokinetics of sodium selenite
* To assess changes in Prostate specific antigen (PSA) To evaluate the anti tumor activity of sodium selenite and abiraterone when given in combination as determined by biochemical progression free survival (PFS) and radiographic PFS.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study. Consent is to be obtained prior to the initiation of any study related tests or procedures that are not part of standard of care for the subject's disease.
* Histologically confirmed adenocarcinoma of the prostate with metastatic disease.
* Progression on abiraterone defined by a rise in PSA at 2 time points at least 1 week apart.
* Male ≥18 years of age.
* Prior orchiectomy or serum testosterone levels < 50 ng/dL determined within 4 weeks prior to start of study drug
* Adequate baseline organ function as defined below:

  * Hemoglobin > 9 with or without transfusion
  * Platelets > 75 with or without transfusion
  * Neutrophil: Absolute neutrophil > 1.0
  * T bilirubin < 1.5 x Upper limit normal (ULN)
  * Aspartate aminotransferase (AST)/Alanine Aminotransferase (ALT) < 2.5 x ULN
  * Creatinine < 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 2 weeks of initiation of study drug administration.
* Ongoing androgen depletion therapy with a gonadotropin releasing hormone (GnRH) analog or inhibitor, or orchiectomy (ie, surgical or medical castration). Note: subjects who have not undergone orchiectomy must continue GnRH analog therapy for the duration of this protocol.
* For subjects previously treated with 1st generation anti androgens (ie, flutamide, nilutamide, or bicalutamide), discontinuation of flutamide or nilutamide therapy must occur > 4 weeks (> 6 weeks for bicalutamide) prior to start of study drug with no evidence of an anti androgen withdrawal response (ie, no decline in serum PSA; within 6 weeks of last dose for bicalutamide and 4 weeks of last dose for all other drugs as above).
* For subjects previously treated with chemotherapy, targeted therapy, immunotherapy, or treatment with an investigational anticancer agent, discontinuation must have occurred ≥ 2 weeks, or after at least 4 half lives, whichever is longer, prior to study drug administration. For enzalutamide and apalutamide, the washout period will be at least 3 weeks prior to start of study drug with no evidence of an anti androgen withdrawal response (ie, no decline in serum PSA within 4 weeks of last dose.)
* For subjects previously treated with other agents approved for the treatment of prostate cancer (5 α reductase inhibitors, estrogens, others), discontinuation of therapy must have occurred ≥ 4 weeks prior to start of study drug. This does not apply to abiraterone.
* Palliative radiotherapy (to bone or soft tissue lesions) must be completed > 2 weeks prior to start of study drug.
* For subjects receiving bone-loss prevention treatment (eg, bisphosphonates or denosumab), the subject must be on stable dose ≥ 4 weeks prior to start of study drug.
* QT interval corrected using Fridericia's method (QTcF) less than 460 msec (see Appendix B for Fridericia's criteria).
* A man who is sexually active with a woman of childbearing potential must agree to use an adequate method of contraception to avoid conception during the study and for 120 days after receiving the last dose of study drug. All men must also not donate sperm during the study and for 120 days after receiving the last dose of study drug.
* Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Previously documented or current brain metastases.
* Untreated spinal cord compression.
* Known positive test result for human immunodeficiency virus.
* History of clinically significant cardiovascular disease including, but not limited to:

  * Myocardial infarction or unstable angina within the 6 months prior to the first dose of study drug.
  * Clinically significant cardiac arrhythmia.
  * Uncontrolled (persistent) hypertension: systolic blood pressure > 180 mHg; diastolic blood pressure >100 mmHg.
  * Congestive heart failure (New York Heart Association class III IV).
* Known active or chronic hepatitis B or hepatitis C as demonstrated by hepatitis B surface antigen positivity and/or anti hepatitis C virus positivity, respectively. Subjects with clinically active or chronic liver disease, including liver cirrhosis of Child Pugh class C, are also excluded.
* History of a different malignancy except for the following circumstances: (a) individuals with a history of other malignancies are eligible if they have been disease free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, (b) individuals with a history of treatment for the following cancers are eligible: non muscle invasive bladder cancer, basal cell, or squamous cell carcinoma of the skin and resected melanoma in situ.
* Any serious underlying medical or psychiatric condition (eg, alcohol or drug abuse), dementia or altered mental status or any issue that would impair the ability of the subject to receive or tolerate the planned treatment, to understand informed consent or that in the opinion of the investigator would contraindicate the subject's participation in the study or that would confound the results of the study.
* Evidence of active viral, bacterial, or systemic fungal infection requiring systemic treatment within 7 days prior to the first dose of study drug. Subjects requiring any systemic antiviral, antifungal, or antibacterial therapy for active infection must have completed treatment no less than 7 days prior to the first dose of study drug.
* Enrollment in another therapeutic study.
* Major surgery (eg, requiring general anesthesia) within 3 weeks before screening, or has not fully recovered from prior surgery (ie, unhealed wound), or surgery planned during the time the subject is expected to participate in the study. Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting Toxicity (DLT) | 2 weeks
  Adverse events will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5. Dose limiting toxicities (DLTs) of the combination of sodium selenite plus abiraterone are defined as:
  * Any ≥ Grade 3 non-hematologic toxicity (possibly, probably, or definitely-related adverse event)
  * Any ≥ Grade 3 thrombocytopenia with bleeding
  * Any ≥ Grade 4 thrombocytopenia persisting > 7 days
  * Any ≥ Grade 4 neutropenia persisting > 7 days
  * Treatment withdrawal by participant decision, or for safety reasons as deemed necessary by the investigator The DLT outcome will be reported as the number of DLT events by dose cohort occurring within 2 weeks of the beginning of treatment, a number without dispersion.

SECONDARY OUTCOMES:
Serious Adverse Events (SAEs | 16 weeks
  Participants will be monitored for 12 weeks of treatment, and for 4 weeks subsequent (up to 16 weeks in total), for serious adverse events. The SAE outcome will be reported as the number of SAEs by dose cohort occurring within 16 weeks of the beginning of treatment, a number without dispersion.
Sodium Selenite Pharmacokinetics | 1 day
  Blood levels of sodium selenite (pharmacokinetics) will be assessed at baseline and through 24 hours after the initial dose. The pharmacokinetics outcome will be reported by dose cohort as the mean blood level with standard deviation
Blood Levels of Prostate-specific Antigen (PSA) | upto 12months
  Maintenance of prostate-specific antigen (PSA) levels in the blood consistent with disease control can be characterized as biochemical progression free survival (PFS). Blood PSA levels will be measured at baseline through treatment. The outcome will be reported as the PSA level by dose cohort at baseline and at the last assessment within 12 months. The values will be reported as the mean with standard deviation.
Radiographic Progression free Survival (PFS) | upto 12months
  Progression free survival (PFS) means continued survival without disease relapse or recurrence. Status will be assessed by regular medical care radiographic scans, eg, computed tomography (CT); positron emission tomography (PET); X-rays; or other scans appropriate for each participant's medical condition, using the last radiographic assessment within 12 months after the start of treatment. Status will be determined per the Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as follows.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in lesion diameters
  * Progressive disease (PD) = 20% increase in lesion diameters, and/or 1+ new lesions
  * Stable disease (SD) = Small changes not meeting above criteria The outcome will be reported by dose cohort as the number of participants remaining alive without disease relapse, progression, or recurrence, a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Knox, Principal Investigator — Stanford Universiy

IPD SHARING:
Plan to Share IPD: No